CLINICAL TRIAL: NCT05808777
Title: Validation of the ICH Score for the Prediction of 12-month Functional Outcome in Patients With Primary Intracerebral Hemorrhage
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201905045RINB
Record Dates: First submitted 2023-03-27; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Intra Cerebral Hemorrhage
Keywords: Intracerebral hemorrhage; Functional outcome; Prognosis; Survivors; Rehabilitation
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICH: Patients were eligible for inclusion if they
  1. were aged 20 years or older
  2. had been admitted to a neurology, neurosurgery, or rehabilitation ward with a diagnosis of primary ICH
  3. had a diagnosis of ICH confirmed by a brain CT
  4. have written informed consent given by themselves or by their legal representative
  Interventions: Other: Phone interview

INTERVENTIONS:
Other: Phone interview — A interview follow-up with a physician by phone was performed at 12 months after the onset of ICH.

SUMMARY:
The goal of this observational study is to analyze the validity of the intracerebral hemorrhage (ICH) Score and a new modified ICH score for the prediction of 12-month functional outcome in patients with primary ICH.

Participants who were admitted to NTUH rehabilitation ward will be followed up to 12 months after the onset of ICH. The follow-up will be conducted by phone interviews.

DETAILED DESCRIPTION:
The ICH Score had been utilized to predict the 30-day mortality after acute intracerebral hemorrhage (ICH), but there's still no reliable tool in predicting the long-term functional outcome in ICH patients. Recently, there have been some studies that use ICH score to predict the prognosis of functional outcome in ICH patients. However, most studies included patients in western societies. Relevant studies in Taiwan were scarce. The present study will follow up the patients with ICH, who were admitted to NTUH rehabilitation ward, up to 12 months post stroke. The follow-up will be conducted by phone interviews at certain time after the onset of ICH. Investigators aim to analyze the validity of the ICH Score for the prediction of 12-month functional outcome in patients with primary ICH. Investigators will also add other variables to see if the revised score could better predict the prognosis among ICH patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years or older
* Had been admitted to a neurology, neurosurgery, or rehabilitation ward with a diagnosis of primary intracerebral hemorrhage (ICH)
* Had a diagnosis of ICH confirmed by a brain computed tomography (CT)
* Have written informed consent given by themselves or by their legal representative

Exclusion Criteria:

* ICH related to aneurysm, arteriovenous malformation, or trauma
* Died before discharge

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A tertiary medical center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Barthel index | 12-month after ICH onset
  Barthel index score, range: 0-100, higher scores mean a better outcome
Modified Rankin scale | 12-month after ICH onset
  Modified Rankin scale, range: 0-6, higher scores mean a worse outcome

SECONDARY OUTCOMES:
Tube retention rate | 12-month after ICH onset
  Including Nasogastric (NG) tube, Foley catheter, tracheal tube
Rehabilitation treatment course | 12-month after ICH onset
  Including inpatient rehabilitation and outpatient rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Mingyen Hsiao, MD, phD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No